CLINICAL TRIAL: NCT03034785
Title: Young Hands at Work and Play: Flexible Electronics for Early Assessment of Force Modulation and Planning in Children Born Prematurely
Brief Title: Flexible Electronics for Early Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyss Institute at Harvard University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Goldfield, Associate Professor of Psychology in Psychiatry, Wyss Institute at Harvard University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: LCD-CS-0001; 1R01HD090985-01 (NIH); IRB16-1008 (Other: Harvard Longwood Medical Area IRB)
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2020-05

CONDITIONS: Very Low Birth Weight Infant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Group 1 (No Intervention): Term
- Group 2 (No Intervention): Preterm
- Group 3 (Experimental): Term
  Interventions: Device: FlexiMitt
- Group 4 (Experimental): Preterm
  Interventions: Device: FlexiMitt

INTERVENTIONS:
Device: FlexiMitt — The proposed research designs and fabricates a new technological innovation in wearable soft-sensors, called flexi-mitts, for measuring force modulation and joint angles of the hand (wrist and fingers) of toddlers.
  Arms: Group 3; Group 4

SUMMARY:
The morbidities associated with very low birth weight (VLBW) infants constitute a major health problem and a significant emotional and financial burden for families and our nation. The key to reducing this burden is early diagnosis. This research will be the first step towards intervention for cerebral growth and long-term neurodevelopmental morbidities of VLBW infants.

The proposed research is to design and fabricate a new technological innovation in wearable soft-sensors, called flexi-mitts, for measuring force modulation and joint angles of the hand (wrist and fingers) of toddlers. Building upon the investigators' ongoing work, they plan to engineer stretchable electronics for safe, toddler-scaled flexi-mitts to measure planning and force modulation.

The investigators' new flexi-mitt technology has the potential to provide a new diagnostic technology and the development of clinical assessment norms. With additional trials of the technology in large numbers of young children, it may be possible for clinicians and day care providers to eventually make measurements of planning and force modulation in play settings.

ELIGIBILITY:
Inclusion Criteria:

Children Born Prematurely ("Preterm") -

Pilot Studies:

* Ages 13-60 months (with the target ages around 18, 24, and 30 months)
* Very low birth weight (less than 1500 grams)
* Born between 28 and 33 weeks
* Parent/Legal guardian provides written consent
* Parent/Legal guardian is willing to facilitate testing with child (and may be included in photos/videos as a result)
* Otherwise healthy condition

Longitudinal Study:

* Ages 13-60 months (with the target age around 24 months) at the time of enrollment
* Very low birth weight (less than 1500 grams)
* Born between 28 and 33 weeks
* Parent/Legal guardian provides written consent
* Parent/Legal guardian is willing to facilitate testing with child (and may be included in photos/videos as a result)
* Otherwise healthy condition

Typically Developing Children ("Term") -

Pilot Studies:

* Ages 13-60 months (with the target ages around 18, 24, and 30 months)
* Born at full term (37 weeks or later)
* Healthy, with no history of neurological problems or musculoskeletal disorders, self-reported by parent or legal guardian
* Parent/Legal guardian provides written consent
* Parent/Legal guardian is willing to facilitate testing with child (and may be included in photos/videos as a result)

Longitudinal Study:

* Ages 13-60 months (with the target age around 24 months) at time of enrollment
* Born at full term (37 weeks or later)
* Healthy, with no history of neurological problems or musculoskeletal disorders, self-reported by parent or legal guardian
* Parent/Legal guardian provides written consent
* Parent/Legal guardian is willing to facilitate testing with child (and may be included in photos/videos as a result)

Exclusion Criteria:

Both Preterm and Term

* Child has a history of/or currently exhibits any severe neurological complications, such as perinatal intraventricular hemorrhage (Grade 3 or 4) or periventricular leukomalacia
* The participant is a child of a PI or other IRB-approved study team member
* Parent/legal guardian does not provide consent or is unwilling to facilitate testing with child

Ages: 13 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Design and Fabricate FlexiMitts | Anticipated Year 1
  To measure joint angles and force
Demonstrate Safety | Anticipated Year 1
  Bench tests of material failure (i.e., stretch deformity and compositional integrity)
Examine group differences between Groups 1 and 2 | Anticipated Year 2 through 4
  To examine group differences in force modulation and joint angles
Examine longitudinal differences between Groups 1 and 2 | Anticipated Year 2 through 4
  To examine longitudinal changes in force modulation and joint angles at 24 and 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Goldfield, Ph.D., Principal Investigator — Wyss Institute for Biologically Inspired Engineering
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wyss Institute for Biologically Inspired Engineering at Harvard University, Boston, Massachusetts

REFERENCES:
- [Background] Lawn JE, Kinney M. Preterm birth: now the leading cause of child death worldwide. Sci Transl Med. 2014 Nov 19;6(263):263ed21. doi: 10.1126/scitranslmed.aaa2563. No abstract available. PMID 25411468
- [Background] Rubens CE, Sadovsky Y, Muglia L, Gravett MG, Lackritz E, Gravett C. Prevention of preterm birth: harnessing science to address the global epidemic. Sci Transl Med. 2014 Nov 12;6(262):262sr5. doi: 10.1126/scitranslmed.3009871. PMID 25391484
- [Background] Back SA. Cerebral white and gray matter injury in newborns: new insights into pathophysiology and management. Clin Perinatol. 2014 Mar;41(1):1-24. doi: 10.1016/j.clp.2013.11.001. PMID 24524444
- [Background] Gordon AM, Duff SV. Fingertip forces during object manipulation in children with hemiplegic cerebral palsy. I: anticipatory scaling. Dev Med Child Neurol. 1999 Mar;41(3):166-75. doi: 10.1017/s0012162299000353. PMID 10210249
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Nordstrand L, Holmefur M, Kits A, Eliasson AC. Improvements in bimanual hand function after baby-CIMT in two-year old children with unilateral cerebral palsy: A retrospective study. Res Dev Disabil. 2015 Jun-Jul;41-42:86-93. doi: 10.1016/j.ridd.2015.05.003. Epub 2015 Jun 19. PMID 26100242
- [Background] Ulrich BD. Opportunities for early intervention based on theory, basic neuroscience, and clinical science. Phys Ther. 2010 Dec;90(12):1868-80. doi: 10.2522/ptj.20100040. Epub 2010 Oct 21. PMID 20966210
- [Background] Adolph KE, Berger SE, Leo AJ. Developmental continuity? Crawling, cruising, and walking. Dev Sci. 2011 Mar;14(2):306-18. doi: 10.1111/j.1467-7687.2010.00981.x. PMID 21399716
- [Background] Goldfield EC, Wolff PH. A dynamical systems perspective on infant action and it's development. Oxford Wiley-Blackwell; 2004
- [Background] Thelen E, Smith L. A dynamic systems approach to the development of cognition and action. Cambridge, MA: MIT Press 1994
- [Background] Slota GP, Latash ML, Zatsiorsky VM. Grip forces during object manipulation: experiment, mathematical model, and validation. Exp Brain Res. 2011 Aug;213(1):125-39. doi: 10.1007/s00221-011-2784-y. Epub 2011 Jul 7. PMID 21735245
- [Background] Santello M, Baud-Bovy G, Jorntell H. Neural bases of hand synergies. Front Comput Neurosci. 2013 Apr 8;7:23. doi: 10.3389/fncom.2013.00023. eCollection 2013. PMID 23579545
- [Background] Eliasson AC, Gordon AM, Forssberg H. Basic co-ordination of manipulative forces of children with cerebral palsy. Dev Med Child Neurol. 1991 Aug;33(8):661-70. doi: 10.1111/j.1469-8749.1991.tb14943.x. PMID 1916022
- [Background] Forssberg H, Eliasson AC, Kinoshita H, Johansson RS, Westling G. Development of human precision grip. I: Basic coordination of force. Exp Brain Res. 1991;85(2):451-7. doi: 10.1007/BF00229422. PMID 1893993
- [Background] Yoshikawa T, Nagai K. Manipulating and grasping forces in manipulation by multifingered robot hands. IEEE Transactions on Robotics and Automation 7:67-77, 1991.
- [Background] Chen YP, Keen R, Rosander K, von Hofsten C. Movement planning reflects skill level and age changes in toddlers. Child Dev. 2010 Nov-Dec;81(6):1846-58. doi: 10.1111/j.1467-8624.2010.01514.x. PMID 21077868
- [Background] Jung WP, Kahrs BA, Lockman JJ. Manual action, fitting, and spatial planning: relating objects by young children. Cognition. 2015 Jan;134:128-39. doi: 10.1016/j.cognition.2014.09.004. Epub 2014 Oct 19. PMID 25460386
- [Background] Park WL, Chen BR, Wood RJ. Design and fabrication of soft artificial skin using embedded micro channels and liquid conductors. IEEE Sensors Journal 12(8):2711-2718, 2012.
- [Background] Park YL, Majidi C, Kramer R, Berard P, Wood RJ. Hyperelastic pressure sensing with a liquid-embedded elastomer. Journal of Micromechanics and Microengineering 20(12), 2010.
- [Background] Majidi C, Kramer R, Wood RJ. A non-differential elastomer curvature sensor for softer-than-skin electronics. Smart Materials and Structures 20(10), 2011
- [Background] Vogt D, Park YL, Wood RJ. Design and characterization of a soft multi-axis force sensor using embedded microfluidic channels. IEEE Sensors Journal 13(10):4056-4064, 2013
- [Background] Endo Y, Tada M, Mochimaru M. Dhaiba: Development of Virtual Ergonomic Assessment System with Human Models Digital Human Modeling 1-8, 2014.
- [Background] Benjamini Y, Hochberg Y. Controlling the false discovery rate: A practical and powerful approach to multiple testing. Journal of the Royal Statistical Society Series B (Methodological) 57(1):289-300, 1995.
- [Background] Diggle P, Liang K-Y, Zeger SL. Analysis of longitudinal data. Clarendon Press; 1994.